CLINICAL TRIAL: NCT04922983
Title: Incobotulinumtoxin A and Yoga-like Isometric Exercise in Adolescent Idiopathic Lumbar Scoliosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manhattan Physical Medicine and Rehabilitation, LLP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00047989
Record Dates: First submitted 2021-04-03; First posted 2021-06-11 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-08

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence; Scoliosis; Lumbar Region
Keywords: Adolescent idiopathic scoliosis; scoliosis; yoga; isometric; botulinum
MeSH Terms: conditions — Scoliosis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Three groups: Group I: Placebo isometric measure, no injection Group II True isometric exercise, placebo injection Group III: True isometric exercise, botulinum injection
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will understand they may receive placebo, and that they will not be told Investigators will know whether they give injections or not, but will not know if injection is placebo.
  Outcomes assessors will be blinded to the entire procedure (radiologists reading X-rays).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I: Placebo isometric measure, no injection (Sham Comparator): Group I: no isometric yoga-like exercise, no injection given.
  Interventions: Behavioral: Placebo
- Group II Isometric yoga-like exercise, placebo injection given (Placebo Comparator): Group II isometric yoga-like exercise, injection of preservative-free normal saline.
  Interventions: Behavioral: Isometric Yoga-like exercise
- Group III: True isometric exercise, botulinum injection (Active Comparator): Group III: Isometric yoga-like exercise, botulinum injection given
  Interventions: Drug: Botulinum toxin type A; Behavioral: Isometric Yoga-like exercise
- Crossover (Active Comparator): After the three months, Arm I and Arm II patients will be given botulinum injections, and Group I will be given the proper yoga-like exercise. These two arms will constitute a further comparator with their own performances in the first 3 months of the study.
  Interventions: Drug: Botulinum toxin type A; Behavioral: Isometric Yoga-like exercise

INTERVENTIONS:
Drug: Botulinum toxin type A — A position similar to the side-plank (Vasisthasana) held for maximal time at least once daily (usual duration: 30 - 90 seconds).
  Other Names: Incobotulinumtoxin A
  Arms: Crossover; Group III: True isometric exercise, botulinum injection
Behavioral: Isometric Yoga-like exercise — Extended torso and legs held diagonally by one straight arm, back against wall if necessary
  Other Names: Side-Plank, Vasisthasana
  Arms: Crossover; Group II Isometric yoga-like exercise, placebo injection given; Group III: True isometric exercise, botulinum injection
Behavioral: Placebo — Used as placebo
  Other Names: no active intervention by drug or yoga-like exercise
  Arms: Group I: Placebo isometric measure, no injection

SUMMARY:
The study uses a yoga-like isometric posture and botulinum injections to reduce the curves in adolescent idiopathic lumbar scoliosis. Three previous studies show that the yoga pose is effective for reversing scoliotic curves; Botulinum toxin has been approved by the FDA for teenagers. However, no studies using the two of them together have been done until this one.

DETAILED DESCRIPTION:
The randomized control 6-month study employs an isometric yoga-like posture to strengthen the weak side, and one set of botulinum injections to weaken the strong side of adolescent idiopathic lumbar scoliosis between 25 and 60 degrees. It is open to people between 12 and 18 years of age who are willing to do the pose every day for three months.

This is a crossover study: After 3 months, every patient who was placebo will be offered the actual proven yoga pose and botulinum toxin injections. Two additional free X-rays at 3 weeks and 3 months following the botulinum injection will also be available to each placebo patient.

In this way every patient - placebo or not - will receive the full proper treatment within 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Fourteen - 18 years of age, 2. Scoliotic curve greater than 25 degrees, less than 45 degrees, 3. Stated willingness to do the yoga and yoga-like poses daily, 4. Written, signed consent by patient and parent/guardian 5. Pre-test Cobb films no less than 3 months old read by independent radiologists.

* Exclusion Criteria:

  1. Neurological, muscular or neuromuscular disease, (e.gs., cerebral palsy, myopathy, stroke),
  2. Genetic abnormalities that affect limb growth, proportionality or metabolism, (e.gs., mucopolysaccharidoses, Marfan's syndrome, Refsums disease).
  3. Pregnancy and other conditions prohibiting X-rays or minute(s)-long exertion (e.gs., congestive heart failure, great weakness, COPD).
  4. Previous exposure to botulinum neurotoxin Type A. Sexually active female subjects must present a recent negative pregnancy test.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in lumbar and thoracic scoliotic curve | At study onset
  Measured by the Cobb angle in coronal X-rays
Reduction in lumbar and thoracic scoliotic curve | 3 weeks after study onset
  Measured by the Cobb angle in coronal X-rays
Reduction in lumbar and thoracic scoliotic curve | 3 months after study onset
  Measured by the Cobb angle in coronal X-rays
Reduction in lumbar and thoracic scoliotic curve | 3 weeks after crossover group injections
  Measured by the Cobb angle in coronal X-rays
Reduction in lumbar and thoracic scoliotic curve | 3 months after crossover group injections
  Measured by the Cobb angle in coronal X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Loren M Fishman, Principal Investigator — Columbia University
Locations (1):
- Manhattan Physical Medicine and Rehabilitation, PLLC, Manhattan, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fishman LM, Groessl EJ, Sherman KJ. Serial case reporting yoga for idiopathic and degenerative scoliosis. Glob Adv Health Med. 2014 Sep;3(5):16-21. doi: 10.7453/gahmj.2013.064. PMID 25568820
- [Result] Fishman LM. Isometric Yoga-Like Maneuvers Improve Adolescent Idiopathic Scoliosis-A Nonrandomized Control Trial. Glob Adv Health Med. 2021 Feb 24;10:2164956120988259. doi: 10.1177/2164956120988259. eCollection 2021. PMID 33717658
- [Result] Fishman LM, Groessl EJ, Bernstein P.Two Isometric Yoga Poses Reduce the Curves in Degenerative and Adolescent Idiopathic Scoliosis. Topics in Geriatric Rehabilitation. 33(4):231-237, October/December, 2017.
- See also: Adult Scoliosis and Yoga Study — https://journals.lww.com/topicsingeriatricrehabilitation/Abstract/2017/10000/Two_Isometric_Yoga_Poses_Reduce_the_Curves_in.3.aspx